CLINICAL TRIAL: NCT04675632
Title: the Director of Vascular Surgery of Hospital of Chengdu University of Traditional Chinese Medicine
Brief Title: Impact of Tibial Run Off on Clinical Outcome of Endovascular Therapy in Femoropopliteal Lesions (TALENT Study)
Status: Completed | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, the director of the vascular surgery of Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCMvs2
Record Dates: First submitted 2020-12-06; First posted 2020-12-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Femoropopliteal Artery Occlusion
Keywords: femoropopliteal artery occlusion; run off score; endovascular therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The intervention group: the tibial run off would be treated through endovascular therapy
  Interventions: Procedure: Endovascular Therapy
- the non-intervention group: the tibial run off would not be treated through endovascular therapy

INTERVENTIONS:
Procedure: Endovascular Therapy — the most commonly used surgical options include: ordinary balloon dilatation， drug-coated balloon (DCB) dilatation and bare stent implantation.
  Groups: The intervention group

SUMMARY:
This study is a prospective, multicenter, real world, observational study intended to understand the impact of tibial run off on clinical outcome of endovascular therapy in Femoropopliteal lesions. It is estimated that 1200 patients with chronic femoral popliteal artery occlusion were enrolled in the group at 8 centers nationwide from January 2021 to December 2022. Two groups would be divided according to whether or not the tibial run off intervened for reconstruction. The intervention group and the non-intervention group. The intervention group would be evaluated Run-off score again after the tibial run off reconstructed. The the Society for Vascular Surgery(SVS) run-off score would be used for the score of the tibial run off. The total score of the tibial run off would be 19 points, 1 point indicating healthy run off. According to the quality of the run off, the preoperative patients would be divided into 1-5, 6-10, 11-15, and >15 points. The follow-up would be conducted at 1, 6, 12, 18 and 24 months after the operation. As it is a real world study, there is no determined end point.The main indicators would be observed including the reintervention rate driven by lesions' clinical symptoms, the rate of primary patency of the femoral popliteal artery, the improvement of quality of life score and rutherford grading.

DETAILED DESCRIPTION:
Arteriosclerosis obliterans of lower extremities (arteriosclerosis obliterans, ASO) is a common and frequently-occurring disease in middle-aged and elderly people, and also an important manifestation of atherosclerosis in lower extremities.ASO is reported to be present in approximately 12%-14% of the population, increasing to 20% of the population over the age of 75.The current treatment methods of ASO include pharmacotherapy, surgical procedures, endovascular treatment, combined surgery, and autologous peripheral blood stem cell transplantation (ASCT), etc.Endovascular treatment of ASO for lower limbs has the advantages of safety, effectiveness and fewer complications, and has become the preferred treatment for ASO.Endovascular treatment mainly includes: percutaneous transluminal angioplasty (PTA) and bare stent implantation. Currently, the most commonly used surgical options include: ordinary balloon dilatation + drug-coated balloon (DCB) dilatation + bare stent implantation.A number of studies have proved that DCB and bare stent are more effective than common PTA, but postoperative restenosis in ASO is always a difficulty.In addition to the chronic total occlusion or diffuse lesion of the lower extremity arteries, the inferior genicular artery outflow channel, age, diabetes, hemodialysis and critical limb ischemia are all related.Matsumi J, et al. found that patency of the inferior genicular artery may be an important predictor of adverse events after the SMART stent implantation in patients with popliteal artery disease, and the preservation of the distal outflow tract may be beneficial to reduce the rate of restenosis Early analysis of the patency rate of inferior genicular artery bypass found that poor outflow tract could lead to an increase in bypass thrombosis events.Matsumi J,et al. found that patency of the Early analysis of the patency rate of inferior genicular artery bypass found that poor outflow tract could lead to an increase in bypass thrombosis events. may be an important predictor of adverse events after SMART stent implantation in patients with popliteal artery disease, and the preservation of the distal outflow tract may be beneficial to reduce the rate of restenosis.Daniel M et al. conducted a retrospective analysis of 95 patients with femoral popliteal artery stent implantation and found that,for patients with poor subgenual artery outflow tract, the number of additional inferior genicular artery during femoral artery stent implantation usually leads to better clinical outcomes.the number of inferior genicular artery shown by preoperative angiography is an independent predictor of post-stent clinical outcomes.This study demonstrates the importance of distal outflow tract clinical outcomes after stent implantation.Yusuke W,et al. conducted a retrospective study on 199 patients with chronic popliteal artery occlusion and found that additional inferior genicular artery opening during stent implantation was beneficial to the patency rate of the stent and clinical results .However, the current analysis of the influence of the tibial run off on the femoral popliteal patency is mainly a retrospective study.

The purpose is to evaluate the patency of the tibial run off through a prospective multicenter observational real world study, whether it has an impact on the therapeutic effect after endovascular treatment in femoral popliteal artery , and whether one-stage reconstruction of the tibial run off can improve the postoperative patency rate of endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Rutherford stages 2-5. 2) The femoral and popliteal artery as the target of the study has at least ≥70% stenosis or occlusion.

  3) Whether it is a primary femoral and popliteal artery disease or in-stent restenosis, patients who received endovascular recanalization successfully (Residual stenosis <30% and no flow-limiting arterial dissection) can be enrolled in the group.

  4) For the patients with both lower limbs to be treated, both limbs can be selected into the group.

  5) Patients who failed the first treatment because the guide wire could not pass through the lesion can still be included in the group after successful endovascular interventional treatment.

  6) Patients who understand the purpose of this research, volunteer to participate in the experiment, sign an informed consent form and are willing to be followed up can be included in the experiment.

  7) For ipsilateral aortoiliac artery disease, patients with residual stenosis <30% can also be included in the group after intravascular reconstruction.

Exclusion Criteria:

* 1) Patients with acute arterial thrombosis. 2) Patients with serum creatinine level> 176μmol/L. 3) Patients with Rutherford stage 5 have foot infection grades of 2 and 3 in the preoperative WIFI (WIfI) classification.

  4) Limbs that have been treated with the femoral and popliteal artery bypass surgery.

  5) Patients who are known to be allergic or sensitive to contrast agents, heparin, aspirin (ASA), other anticoagulant or antiplatelet therapies, and/or paclitaxel.

  6) Patients with bleeding constitution. 7) Pregnant and lactating women. 8) Patients with a history of myocardial infarction or unstable angina within 3 months.

  9) Patients with a history of TIA or cerebral infarction within 3 months. 10) Patients with severe disease such as liver failure. 11) Patients with a life expectancy of less than 24 months. 12) Participating in other drug or device studies currently. 13) Patients with poor treatment compliance or deemed unsuitable for inclusion in the group by the researcher.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Arteriosclerosis obliterans of lower extremities
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
the clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 24 months
  Any reintervention within the target lesion due to symptoms or drop of ABI≥20% or >0.15 when compared to post-index procedure baseline ABI.
Changes of the patency rate of target(Femoropopliteal) lesions at post-interventional | baseline and 24 months
  the patency rate of target(Femoropopliteal) lesions would be determined by vascular ultrasound,Restenosis would be diagnosed if the peak systolic velocity ratio(PSVR)≥2. 5.

SECONDARY OUTCOMES:
vascular quality of life questionnaire(VascuQol) | 1 month,6 months,12 months,18 months and 24 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Wound,Ischemia,and foot infection(WIFI) classification system | 1 month,6 months,12 months,18 months and 24 months
  The Wound, Ischemia, and foot Infection (WIfI) classification system was created to encompass demographic changes and expanding techniques of revascularization to perform meaningful analyses of outcomes in the treatment of the threatened limb,including wound,ischemia and foot infection.Each index was evaluated by very low,low,moderate and high,the very low represents no risk,the high reveals high risk of amputation.
Changes of rutherford grade | 1 month,6 months,12 months,18 months and 24 months
  Rutherford classified Peripheral arterial disease(PAD) into acute and chronic limb ischemia, emphasizing that each presentation requires different treatment algorithms.The system was based on clinical symptoms and objective findings, including Doppler, arterial brachial indices (ABI), and pulse volume recordings.Rutherford's acute limb ischemia(ALI) classification divides an extremity into viable, threatened, or irreversibly damaged categories from 0-6,the lowest reveals no hemodynamically significant occlusive disease,the highest shows functional foot no longer salvageable.
Incidence of perioperative adverse events | 1 month,6 months,12 months,18 months and 24 months
  To measure the safety of the whole procedure,adverse events including acute vascular event,major adverse events related to surgery(major amputation,death) wound be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, doctor, Principal Investigator — RenJi Hospital; Ziheng Wu, doctor, Principal Investigator — Zhejiang University; Lianrui Guo, doctor, Principal Investigator — Xuanwu Hospital, Beijing; Xin Fang, doctor, Principal Investigator — Hangzhou First People's hospital of Medical College of Zhejiang University; Hongfei Sang, doctor, Principal Investigator — Second Affiliated Hospital of Suzhou University; Zibo Feng, doctor, Principal Investigator — Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology; Qiang Li, doctor, Principal Investigator — Qingdao Haici Hospital
Locations (1):
- Chunshuihe, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Liu Y, Wang Q, Wu Z, Fen Z, Guo L, Li Q, Fang X, Sang H, Dai Y, He C, Ye M. A prospective, multicenter, real-world observational study evaluating the impact of tibial runoff on clinical outcomes after endovascular therapy for femoropopliteal lesions: Research protocol. Front Cardiovasc Med. 2022 Nov 16;9:1035659. doi: 10.3389/fcvm.2022.1035659. eCollection 2022. PMID 36465469